CLINICAL TRIAL: NCT06388720
Title: A Study to Assess the Clinical Effectiveness and Safety of Intravesical Mitomycin-C and Gemcitabine Sequential Therapy in Patients With High Risk Non-muscle Invasive Bladder Cancer (NMIBC) Unresponsive to BCG Therapy
Brief Title: The Clinical Effectiveness and Safety of Intravesical Mitomycin-C and Gemcitabine Sequential Therapy
Acronym: IMGeS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Ho Kyung Seo, Primary Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2024-0026
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-05

CONDITIONS: Bladder Cancer
Keywords: high risks non-muscle invasive bladder cancer; Sequential treatment; Intravesical treatment; Mitomycin-c; Gemcitanine
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Mitomycin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Intravesical sequential treatment of Mitomycin-c 40mg/20ml and Gemcitabine 2000mg/50ml
  Interventions: Drug: Mitomycin-C; Drug: gemcitabine

INTERVENTIONS:
Drug: Mitomycin-C — Intravesical instillation of Mitomycin-c 40 mg in 20 ml as the first agent in sequential treatment.
  Other Names: Sequential treatment group
Drug: gemcitabine — Intravesical instillation of Gemcitabine 2000 mg in 50 ml following Mitomycin-c administration.

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of mitomycin-c and gemcitabine sequential instillation in BCG unresponsive high risk non-muscle invasive bladder cancer patients.

DETAILED DESCRIPTION:
Phase 2 clinical, multi-institutional, open assignment prospective study

Primary Outcome Measures:

1-year recurrence-free survival period in high-risk groups after sequential injection of Mitomycin-c 40 mg/20 ml and Gemcitabine 2000 mg/50 ml in non-muscle invasive bladder cancer patients in BCG-free high-risk groups.

Secondary Outcome Measures:

Progression Free Survival (PFS), Cystectomy free survival (CFS), Cancer specific survival (CSS), Overall survival (OS) and safety after Mitomycin-c 40mg/20ml and Gemcitabine 2000mg/50ml treatment in non-muscle invasive bladder cancer patients in BCG-free high-risk groups.

ELIGIBILITY:
Inclusion Criteria:

1. a patient over the age of 20
2. Patients who are willing and able to complete a written test subject consent/approval for this examination.
3. Patients with histological confirmation of high-risk non-muscle infiltration (T1, high-grade Ta and/or CIS) bladder transition cell cancer. However, according to the definition of EAU guidelines high-risk NMIBC, Ta, low grade, and multiple recurrences of more than 3 cm are included.
4. The most recent bladder examination/TURBT must be performed within 8 weeks before the initial administration of the trial treatment. Patients with high risk NMIBC who received proper BCG treatment but did not respond to BCG
5. Patients who are not eligible for a radical bladder resection or who have refused surgery.
6. Patient who are not being pregnant or breast feeding until the study period.

Exclusion Criteria:

1. Patient diagnosed with muscle-invasive bladder cancer at TURBT
2. If upper urinary tract urothelial cancer is accompanied by imaging
3. If the imaging indicates extravesical involvement (cT3)
4. Imaging shows lymph node metastasis (short-axis 15mm or more) or distant metastasis
5. In a biopsy, non-transitional cell histology is dominant, or only non-transitional cell tissue is present (primary squamous cell carcinoma, primary adenocarcinoma, small cell carcinoma, sarcoma, carcinosarcoma, paraganglioma, melanoma, lymphoma)
6. In the case of receiving systemic cytotoxic chemotherapy for other cancers within 3 years
7. If patient have a history of pelvic radiation therapy for other cancers within 3 years
8. If patient have a history of receiving Mitomycin-c or gemcitabine in the bladder within 3 years. The exception is cases used for the purpose of injection therapy of anticancer drugs in the early bladder cancer
9. If patient has a history of allergy to mitomycin-c or gemcitabine
10. Cystoscopy shows a tumor in the prostate urethra
11. Patients who have participated in studies using clinical trial drugs and are currently receiving clinical trial drugs or who have used clinical trial drugs or clinical trial medical devices within 4 weeks prior to the date of initial treatment
12. After post-cystoscopy/TURBT, the patient received intravesical chemotherapy prior to the start of trial treatment
13. Thrombocytopenia, coagulopathy or bleeding tendency patient.
14. Pregnant or breast-feeding women
15. If patient treated yellow fever vaccine or phenytoin
16. Dysfunction of liver or kidney (GFP≤30)
17. If patient undergo severe myelosuppression
18. If patient complicated severe infection
19. If patient definitely diagnosed interstitial lung disease or lung fibrosis by chest X-ray.
20. If patient conduct chest radiotherapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
High risk Recurrent free survival in sequential treatment group. | 1year
  Time from initial TURBT* to first histologically confirmed recurrence of high-risk NMIBC or disease progression (per PFS definition), whichever occurs first.

SECONDARY OUTCOMES:
Progression free survival in sequential treatment group. | 1year
  defined as the period from the initial TURBT date* to the time when T stage progresses (e.g., Ta>T1, CIS>T1) (PFS1) or muscle invasive bladder cancer (T2 or higher) was first biopsy confirmed (PFS2) or imagingally diagnosed with metastasis to bladder cancer.
Cystectomy free survival in sequential treatment group. | 1year
  Defined as the period from the initial TURBT date* to the time when radical cystomy was performed.
cancer specific survival in sequential treatment group. | 1year
  Duration from initial TURBT date* to the time of death from bladder cancer
Overall survival in sequential treatment group. | 1year
  The period from the initial TURBT date* to the point of death (regardless of cause)
Safety of sequential treatment. | 2year
  The first safety analysis is conducted on test subjects who have developed toxicity in accordance with CTCAE standards. In particular, urinary disorders such as urinary tract infections and acute urination that occurred after injection of drugs into the bladder are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Kyung Seo, MD, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, South Korea

IPD SHARING:
Plan to Share IPD: No